CLINICAL TRIAL: NCT01793311
Title: The Effect of Dosage of Caffeine on Intraocular Pressure in Healthy Subjects
Brief Title: The Effect of Dosage of Caffeine on Intraocular Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Damrong Wiwatwongwana, M.D., Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OPT-11-03-03A-12-X
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Intraocular Pressure; Caffeine Dosage
Keywords: intraocular pressure; caffeine; dosage
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group1: Decaffeinated coffee (Sham Comparator): contains 0.5-2 mg of caffeine
  Interventions: Other: decaffeinated coffee
- Group2: regular dose coffee (Active Comparator): contains 91.8 mg of caffeine
  Interventions: Other: regular dose coffee
- Group3: high dose coffee (Active Comparator): contains 144 mg of caffeine
  Interventions: Other: high dose coffee

INTERVENTIONS:
Other: decaffeinated coffee — contains caffeine 0.5-2 mg
  Arms: Group1: Decaffeinated coffee
Other: regular dose coffee — contains 91.8 mg of caffeine
  Arms: Group2: regular dose coffee
Other: high dose coffee — contains 144 mg of caffeine
  Arms: Group3: high dose coffee

SUMMARY:
The goal of the study is to determine the effect of different doses of caffeine on intraocular pressure. We hypothesized that higher dosage of caffeine would increase intraocular pressure more than lower doses.

Eligible subjects will be randomized into three groups:

1. group 1: intake of decaffeinated coffee
2. group 2: intake of coffee with lower caffeine dose
3. group 3: intake of coffee with higher caffeine dose

Intraocular pressure will be measured at 0, 30, 60 and 90 minutes after coffee intake.

DETAILED DESCRIPTION:
decaffeinated coffee contains 0.5-2 mg of caffeine regular dose coffee contains 91.8 mg of caffeine high dose coffee contains 144 mg of caffeine

all three groups' intraocular pressure will be measured with the Goldmann applanation tonometer at 4 timepoints:

1. 0 minutes (baseline)
2. 30 minutes after intake
3. 60 minutes after intake
4. 90 minutes after intake

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* normal central corneal thickness
* normal baseline intraocular pressure

Exclusion Criteria:

* any ocular disease
* baseline intraocular pressure over 21 mmHg
* central corneal thickness less than 520 microns or more than 540 microns

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
change from baseline in intraocular pressure (mmHg)after caffeine intake | 0, 30 minutes, 60 minutes, 90 minutes post-caffeine intake
  intraocular pressure measured at 4 timepoints:
  1. 0 minutes (baseline)
  2. 30 minutes after intake
  3. 60 minutes after intake
  4. 90 minutes after intake

CONTACTS AND LOCATIONS:
Overall Officials: Damrong Wiwatwongwana, M.D., Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University Hospital, Muang, Chiang Mai, Thailand